CLINICAL TRIAL: NCT05587985
Title: The Effect of Early Mobilization on Pain and Mobility Levels in Patients Undergoing Total Knee Prothesis
Brief Title: The Effect of Early Mobilization on Pain and Mobility Levels
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Bartın Unıversity (Other)
Responsible Party: Principal Investigator, Mediha Didem Kocoglu Agca, Research Assistant, Bartın Unıversity
Other Study IDs: 2022-SBB-0345
Record Dates: First submitted 2022-10-06; First posted 2022-10-20 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Early Ambulation
Keywords: Total knee replacement; early mobilization; pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental Group: * After randomization, 34 patients will be included in the experimental group. This group is the group to be mobilized early after surgery.
  * During the data collection process, the pain level of the experimental group will be evaluated at the 8th hour after the operation, then the level of mobility will be evaluated by providing mobilization.
  * At the 20th hour after the surgery, pain assessment of both groups will be made, and then their mobility will be evaluated, and their mobility levels will be evaluated.
- Control Group: * After randomization, 34 patients will be included in the control group. This group is the group that did not undergo early mobilization.
  * The control group will only be evaluated for pain at the 8th hour after surgery, and they will not be mobilized.
  * At the 20th hour after the surgery, pain assessment of both groups will be made, and then their mobility will be evaluated, and their mobility levels will be evaluated.

SUMMARY:
Objective: This study will be conducted to determine the effect of early mobilization on pain and mobility levels in patients who underwent total knee prothesis.

Method: This study, which was designed as a randomized controlled experimental type, will be conducted with a total of 68 patients, 34 of whom were in the control group and 34 in the experimental group, who underwent total knee prothesis surgery in the orthopedics and traumatology service at Bartın State Hospital between September 2022 and June 2023. Research data will be collected with Participant Information Form, Brief Pain Inventory, Patient Mobility Scale and Observer Mobility Scale. During the data collection process, the pain level of the experimental group will be evaluated at the 8th hour after the operation, then the level of mobility will be evaluated by providing mobilization. The control group will only be evaluated for pain at the 8th hour after surgery, and they will not be mobilized. At the 20th hour after the surgery, pain assessment of both groups will be made, and then their mobility will be evaluated, and their mobility levels will be evaluated. SPSS 22.0 program will be used in the evaluation of the data. Whether the data is normally distributed or not will be tested by Shapiro-wilk analysis. According to the result of this, parametric and nonparametric methods will be used.

DETAILED DESCRIPTION:
Introduction: Pain development is an expected situation in individuals who have undergone total knee replacement surgery. Again, in these patients, the tendency to stay still increases due to the surgery and pain. International guidelines and other studies indicate that early mobilization of patients after surgical interventions is effective in preventing complications that can be caused by inactivity and reducing the severity of pain in patients. Early mobilization gains importance in order to accelerate the recovery process of patients after total knee replacement surgery and to prevent problems such as muscle mass loss and muscle weakness that may arise from long-term bed rest.

Objective: This study will be conducted to determine the effect of early mobilization on pain and mobility levels in patients who underwent total knee replacement.

Method: This study, which was designed as a randomized controlled experimental type, will be conducted with a total of 68 patients, 34 of whom were in the control group and 34 in the experimental group, who underwent total knee replacement surgery in the orthopedics and traumatology service at Bartın State Hospital between September 2022 and June 2023. Research data will be collected with Participant Information Form, Brief Pain Inventory, Patient Mobility Scale and Observer Mobility Scale. The patients in the experimental group will not be mobilized until the 8th hour, and their first mobilization will be carried out at the 8th hour. The pain levels of the patients in the experimental group at the 8th hour will be evaluated with the Brief Pain Inventory and their mobilization will be ensured. Mobility levels after mobilization will be recorded by evaluating with the Patient Mobility Scale and by the research nurse who mobilized the patient with the Observer Mobility Scale. Patients in the control group will not be mobilized until the 20th hour after surgery. Patients will be evaluated only for pain at the 8th hour after surgery. The first mobilizations will be made at the 20th hour after the surgery, and their mobility levels will be evaluated with the Observer Mobility Scale and the Patient Mobility Scale by both the patient and the researching nurse who mobilized them. Pain assessment will be performed in both groups at the 20th hour and then their mobility will be evaluated. SPSS 22.0 program will be used in the evaluation of the data. Whether the data is normally distributed or not will be tested by Shapiro-wilk analysis. According to the result of this, parametric and nonparametric methods will be used.

Conclusion: If the research is carried out successfully, the differences caused by early mobilization in the pain levels and mobility levels of the patients will be revealed. The fact that early mobilization causes a decrease in the level of pain, as stated in the literature, will enable patients to be mobilized earlier. Again, if early mobilization has a positive effect on the mobility level of the patients, the patients will be able to be mobilized early for this purpose.

ELIGIBILITY:
Inclusion Criteria:

* Having a total knee replacement surgery
* Volunteering
* Being over 18 years old

Exclusion Criteria:

* Not volunteering
* Patients for whom early mobilization is contraindicated (without physician approval)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients who were hospitalized in the orthopedics and traumatology service of Bartın State Hospital and who had undergone total knee replacement surgery constitute the scope of this study.
Sampling Method: Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
pain status | 8 hours
  At the 8th hour, the pain status of the patients in the control and experimental groups will be evaluated with the Brief Pain Inventory.
  Brief Pain Inventory; It is a form consisting of 9 questions in total. The first question compares the individual's pain with past pain experiences, the second question includes an image where the individual will mark the pain area. The next four questions serve to measure pain intensity with a numerical pain scale. Numerical pain scale is evaluated in the range of 0-10. "0" means no pain, "10" means unbearable pain. The last question evaluates the level of influence of factors such as mobility, emotional state, breathing, coughing exercise, interpersonal relations, walking, working and enjoying life, sleep, due to pain in the last 24 hours, with a value in the range of 0-10. "0" means not affected at all, "10" means completely affected. The higher the score, the higher the pain intensity.
level of mobility | 8 hours
  At the 8th hour, the mobility levels of the patients in the control and experimental groups will be evaluated with the Observer Mobility Scale.
  Observer Mobility Scale: While performing four activities after surgery, dependency/independence status and degree are evaluated between 1 and 5. 1 indicates that the patient cannot perform the activity independently without the need for verbal stimulation or physical assistance, and 5 indicates that the patient cannot perform the activity even with verbal stimulation or physical assistance. As a result, the Global Patient Mobility score is obtained by summing the scores of all activities. The minimum and maximum score that can be obtained from the scale is between 1-5, and the total score is between 4-20. An increase in the score indicates that the patient's mobility skills are insufficient, and a decrease in the score indicates that the patient's mobility is sufficient after the surgery.
pain status | 20 hours
  At the 20th hour, the pain status of the patients in the control and experimental groups will be evaluated with the Brief Pain Inventory.
  Brief Pain Inventory; It is a form consisting of 9 questions in total. The first question compares the individual's pain with past pain experiences, the second question includes an image where the individual will mark the pain area. The next four questions serve to measure pain intensity with a numerical pain scale. Numerical pain scale is evaluated in the range of 0-10. "0" means no pain, "10" means unbearable pain. The last question evaluates the level of influence of factors such as mobility, emotional state, breathing, coughing exercise, interpersonal relations, walking, working and enjoying life, sleep, due to pain in the last 24 hours, with a value in the range of 0-10. "0" means not affected at all, "10" means completely affected. The higher the score, the higher the pain intensity.
level of mobility | 20 hours
  At the 20th hour, the mobility levels of the patients in the control and experimental groups will be evaluated with the Patient Mobility Scale.
  Patient Mobility Scale: It is applied to evaluate the level of pain and difficulty in performing the four activities: turning from one side to the other in the bed, sitting by the bed, standing up by the bed and walking in the patient's room after the surgery. The numerical value of the degree of pain and difficulty is determined by measuring the distance between the mark on the scale and zero with a calibrated ruler. There are two subgroup questions for each activity. The questions are answered as 1 to 5 to determine the level and severity of pain perception, 1 was no pain, 5 was the worst pain I could imagine, and the difficulty levels of the activities were between 1 and 5, 1 was very easy, 5 was very difficult. As a result, the Global Patient Mobility score is obtained by summing the scores of all activities.

SECONDARY OUTCOMES:
pain levels | 0-20 hours
  The correlation between the sociodemographic and clinical characteristics of the patients (patient's age, gender, educational status, height, weight, BMI, analgesic drug used, anesthesia method applied during the operation and duration of the operation) in the experimental and control groups and their pain status will be evaluated with the Brief Pain Inventory at the 8th and 20th hours.
  Brief Pain Inventory; It is a form consisting of 9 questions in total. The first question compares the individual's pain with past pain experiences, the second question includes an image where the individual will mark the pain area. The next four questions serve to measure pain intensity with a numerical pain scale. Numerical pain scale is evaluated in the range of 0-10. "0" means no pain, "10" means unbearable pain. The last question evaluates the level of influence of factors such as mobility, emotional state, breathing, coughing exercise, interpersonal relations, walking, working and enjoying life,
mobility levels | 0-20 hours
  The correlation between sociodemographic and clinical characteristics of the patients (patient's age, gender, educational status, height, weight, BMI, analgesic drug used, anesthesia method applied during the operation and duration of the operation) in the experimental and control groups and their the Observer Mobility Scale and the Patient Mobility Scale will be evaluated with at the 8th and 20th hours.
  Patient Mobility Scale: It is applied to evaluate the level of pain and difficulty in performing the four activities: turning from one side to the other in the bed, sitting by the bed, standing up by the bed and walking in the patient's room after the surgery. The numerical value of the degree of pain and difficulty is determined by measuring the distance between the mark on the scale and zero with a calibrated ruler. There are two subgroup questions for each activity. The questions are answered as 1 to 5 to determine the level and severity of pain perception.

CONTACTS AND LOCATIONS:
Overall Officials: Mediha Didem KOCOGLU, Study Chair — Bartın Unıversity